CLINICAL TRIAL: NCT05651334
Title: Transcranial Magnetic Stimulation in Smokers: an Examination of Mediating Neural Pathways.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kent State University (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, William Lechner. PhD, Assistant Professor, Kent State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-604
Record Dates: First submitted 2022-11-28; First posted 2022-12-15 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to active or sham transcranial magnetic stimulation. Assignment to condition will be conducted using the Urn randomization procedure to ensure balancing on nicotine dependence, and age.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Condition assignment using the URN procedure will be conducted by the research coordinator who is not involved in treatment delivery or outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active repetitive Transcranial Magnetic Stimulation (rTMS) (Experimental): rTMS will be delivered with a MagPro R-30 magnetic stimulator (MagVenture, Farum, Denmark) Cool-B65 A/P (Active/Placebo). Participants will receive 900 pulses of 20 Hz rTMS per session at 110% of the Motor threshold (MT) (45 20-pulse trains of 1 second duration with an inter-train interval of 20 seconds). MT will be established to determine the intensity of stimulation for each participant, as recommended by safety guidelines. MT will be defined as the amount of energy required to induce a visible twitch in contralateral hand in at least 50% of stimulations. The target stimulation site will be the left DLPFC, specifically: located 6 cm anterior of the MT site identified with assistance from the neuro-navigation system to ensure that the target is located in the middle of the frontal gyrus, in the lateral part of Brodmann Area (BA) 9, near the border of BA 46.
  Interventions: Device: Active repetitive Transcranial Magnetic Stimulation
- Sham repetitive Transcranial Magnetic Stimulation (rTMS) (Sham Comparator): Sham rTMS will appear identical to active treatment, with the exception that the sham side of the coil will be used resulting in no stimulation being applied to the participant, while providing a sensation of stimulation.
  Interventions: Device: Sham repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Active repetitive Transcranial Magnetic Stimulation — Active stimulation
  Arms: Active repetitive Transcranial Magnetic Stimulation (rTMS)
Device: Sham repetitive Transcranial Magnetic Stimulation — Sham stimulation
  Arms: Sham repetitive Transcranial Magnetic Stimulation (rTMS)

SUMMARY:
The primary objective of this study is to examine the effects of repetitive transcranial magnetic stimulation (rTMS) on a regulation of craving task (ROC task) and evaluate the feasibility of targeting rTMS via fMRI based neuronavigation. Specifically, we will examine BOLD activation within the DLPFC when control over craving is exerted in order to identify if 1) the task produces reliable activations in an area capable of being targeted by a standard figure-8 coil and 2) examine if the coordinates of the area are distinct from the area targeted via anatomical neuronavigation alone. Last, we will examine if rTMS, compared to sham, is capable of improving cognitive control over craving measured at outcome. The current pilot study will examine these aims in a sample of tobacco dependent adults (N=16) (with final sample size dependent on availability of funds).

DETAILED DESCRIPTION:
The study will include functional magnetic resonance imaging at baseline as well as demographic, psychological, and tobacco use assessments. Following initial assessment, participants will undergo one active rTMS session (20 Hz rTMS, 900 pulses per session, applied to left DLPFC). The outcome session will include assessments repeated from baseline.

The current proposal will examine the following aims. Aim 1: To test the potential for active rTMS to improve cognitive control of craving. Hypothesis: Active rTMS (compared to sham rTMS) will result in significant improvement in control over craving assessed by self-reported craving during the ROC task as well as in terms of activity in prefrontal regions associated with cognitive control during the ROC task.

Aim 2 (feasibility): To examine the feasibility of using fMRI BOLD activation in the DLPFC during the ROC task to target rTMS. BOLD activations during successful control over craving trials will be examined in terms of their reliability within participant and their feasibility as a target for rTMS delivered via standard figure 8 coil (capable of inducing synaptic firing 1.5-3.0 cm beneath the scalp). Additionally, the coordinates for the target identified via BOLD activation during the ROC task will be compared to the coordinates for the target identified by using standard neuronavigation to the DLPFC via anatomical fMRI, in order to determine if these areas are distinct in terms of the direct effect of the stimulation field (approximately 5 cm2).

ELIGIBILITY:
Inclusion Criteria:

* Smokers endorsing atleast moderate dependence (total Fagerstrom for Cigarette Dependence score > 4)
* Endorsing no specific plan to quit smoking in the next 3 months.
* Must meet safety guidelines for application of rTMS
* 18-60 years of age
* Smoked cigarettes regularly for at least one year
* Currently smoke at least 10 cigarettes per day
* Have a carbon monoxide (CO) level greater or equal to 10 ppm
* Currently be using no other nicotine products.

Exclusion Criteria:

* Subjects will be excluded if they meet criteria for current alcohol (moderate - severe), current substance dependence, current affective disorder (depression, dysthymia, or mania) or current psychotic symptoms as assessed by the (MINI) International Neuropsychiatric Exam
* Are currently pregnant or lactating, or intend to become pregnant
* Have a health condition for which rTMS is contraindicated
* Submit a urine drug screen positive for illicit substances or substance misuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Regulation of Craving Task | Assessed during the baseline session and repeated at the outcome session (following stimulation), occurring on average less than one month apart. Primary outcome measure are the ratings collected at the final outcome session.
  Self report ratings of cue induced craving for smoking after instruction. Specifically, differences in craving following positive vs. negative instructions will be compared between active stimulation and sham stimulation groups at the final outcome session, accounting for baseline values (similar to methods detailed in (Kober, Kross, Mischel, Hart, & Ochsner, 2010).
  Kober, H., Kross, E. F., Mischel, W., Hart, C. L., & Ochsner, K. N. (2010). Regulation of craving by cognitive strategies in cigarette smokers. Drug and Alcohol Dependence, 106(1), 52-55. doi:10.1016/j.drugalcdep.2009.07.017
Brief Questionnaire of Smoking Urges (QSU - Brief) | Assessed during the baseline session and repeated at the outcome session (following stimulation), occurring on average less than one month apart. Primary outcome measure are the ratings collected at the final outcome session.
  Self report assessment smoking urges will be compared between active stimulation and sham stimulation groups at the final outcome session, accounting for baseline values.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
NO IPD will be shared.